CLINICAL TRIAL: NCT03235895
Title: Evaluation of Internet-Based CME for Wet-cupping Providers: Randomized Controlled Trial
Brief Title: Evaluation of Internet-Based CME for Wet-cupping Providers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Center for Complementary and Alternative Medicine, Saudi Arabia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: nccam_1_2017
Record Dates: First submitted 2017-07-23; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet based (Experimental): * Six days of Instructional online CME educational material using Test-Enhanced E-Learning strategy.
  * Followed by one day face to face CME activity
  Interventions: Other: Educational material
- Face to Face (Active Comparator): Three days face to face Conventional CME educational materials
  Interventions: Other: Educational material
- Wait listed (No Intervention): No CME activity will be given

INTERVENTIONS:
Other: Educational material — Educational material given as a part of CME activity as through enhanced internet method
  Other Names: CME
  Arms: Face to Face; Internet based

SUMMARY:
A randomized controlled Trial to evaluate the internet based CME for wet cupping providers in Saudi Arabia

DETAILED DESCRIPTION:
Research problem:

Complementary and Alternative Medicine (CAM) is widely used in Saudi Arabia. As wet-cupping practice regulation and licensing had been established the need increased to develop a system of Continuing Medical Education (CME) for wet-cupping providers. E-learning grown steadily to become a popular approach in medical education with the fast-evolving technologies made it possible to develop and implement a high-quality Internet-based CME. The aim of this study is to compare the effectiveness of Internet-based CME with conventional CME in the field of complementary medicine.

Research Significance:

Aiming to control the training to guarantee evidenced-based quality care while facing the challenge of increased number of licensed cupping providers who needs CME hours to maintain and improve their practice. There is a need for a study to evaluate if the internet-based technique can help overcome the challenge and to increase the number and improve the quality of CME activities.

Research Objectives:

To evaluate the effect of internet-based CME activity on knowledge, knowledge retention and intellectual skills in wet-cupping providers compared with conventional CME activity. Moreover, to develop a model of a blended CME activity using the online platform to conduct a flipping classroom CME activity in complementary medicine.

Research Methodology:

Randomised, open, comparative controlled trial. Participants will be selected from a list of the registered cupping providers. Using a list of registered cupping providers (sample frame) a sample will be selected randomly using computer generated number. After taking informed consent participants will be allocated randomly into three groups; 1) Internet-based CME activity group; 2) Conventional CME activity group, and 3) control group (waitlist) receiving no intervention. Data will be explored for distribution, and the appropriate methods of presentation and testing of differences will be selected accordingly. Two-tailed values of p<0.05 will be considered statistically significant. Immediate knowledge score, Retention Knowledge rate and skills score will be compared within and between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, nurses, physiotherapists
* Passed the Compulsory wet cupping training course within the last three years.
* Available during the study periods.

Exclusion Criteria:

* Unaccredited wet cupping training courses.
* Accredit courses more than three Years

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-09-25 (Estimated); Primary Completion 2017-11-25 (Estimated); Study Completion 2017-12-10 (Estimated)

PRIMARY OUTCOMES:
Knowledge score | Day 0 and day 7
  To measure the change the knowledge score within and between the internet-based CME group, the conventional CME group, and the control group before and immediately after the intervention

SECONDARY OUTCOMES:
Knowledge score | Day 7 and day 14
  to asses the change in knowledge score knowledge between day 7 and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Moahmed Khalil, MD, Study Chair — National Center for Complmentary and Alternative Medicine; Abdullah AlMudiaheem, MBBS, Principal Investigator — National Center for Complmentary and Alternative Medicine; Nasser Al-Hamdan, Study Director — College of Medicine

IPD SHARING:
Plan to Share IPD: No